CLINICAL TRIAL: NCT06392334
Title: The Role of Mast Cells and Its Proteases in Chronic Obstructive Pulmonary Disease
Brief Title: Mast Cells and Its Proteases in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Voronezh N.N. Burdenko State Medical Academy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Voronezhsma
Record Dates: First submitted 2019-09-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: COPD Exacerbation
Keywords: mast cell; tryptase; chymase; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy (Other): Biopsy of lung tissue will be done
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Biopsy of lung tissue

SUMMARY:
Mast cells proteases such as chymase and tryptase will be studied in the tissue of small and large airways in COPD patients

ELIGIBILITY:
Inclusion Criteria:

- COPD patients

Exclusion Criteria:

Other lung diseases, tumors, pregnancy

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of mast cells in COPD lung tissue | up to 10 -12 months
  Assesment of mast cells in lung tissue in COPD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Voronezh State Medical University, Voronezh, Russia

IPD SHARING:
Plan to Share IPD: No